CLINICAL TRIAL: NCT00240162
Title: A Phase II Study of PTK787/ZK 222584, a Novel, Oral Angiogenesis Inhibitor as Post Transplant Maintenance Therapy in Patients With Multiple Myeloma Following High Dose Chemotherapy and Autologous Stem Cell Transplant
Brief Title: PTK/ZK as Post Transplant Maintenance Therapy in Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: investigator letter from drug manufacturer stating animal studies showed increased risk of cancer which was an unknown adverse event
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-0639; IND#: 72,721
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Results first posted 2014-09-04 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; PTK
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — vatalanib

ARMS (1):
- PTK787/ZK 222584 (Experimental): Initially patients will receive a dose of 500mg (2, 250mg tablets) in the morning and 250mg (1, 250mg tablet) in the afternoon for 2 weeks (cycle 1, days 1-14), then 500mg (2, 250mg tablets) bid for 2 weeks (cycle 1, days 15-28) and finally 750mg (3, 250mg tablets) in the morning and 500mg (2, 250mg tablets) in the afternoon for the remainder of treatment duration (cycle 2, day 1 and onwards). Each 28 days of drug administration will constitute one cycle of therapy.
  Interventions: Drug: PTK787/ZK 222584

INTERVENTIONS:
Drug: PTK787/ZK 222584
  Other Names: N/Bemzoylstaurosporine

SUMMARY:
The purpose of this study it to evaluate the efficacy of PTK787/ZK 222584, in inducing at least a 50% reduction in paraprotein in patients with multiple myeloma whose paraprotein levels are < 5 g/dL following high dose chemotherapy (HDCT) and autologous stem cell transplantation (ASCT).

DETAILED DESCRIPTION:
To evaluate the efficacy of PTK787/ZK 222584, in inducing at least a 50% reduction in paraprotein in patients with multiple myeloma whose paraprotein levels are < 5 g/dL following high dose chemotherapy (HDCT) and Autologous Stem Cell Transplantation (ASCT).

To assess the time to progression and disease free survival of patients treated with PTK787/ZK 222584.

To assess the safety and tolerability of PTK787/ZK 222584 in multiple myeloma patients following ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for this trial are those diagnosed with multiple myeloma by standard criteria and treated with HDCT and ASCT on protocols at Washington University School of Medicine. Following HDCT and ASCT patients must have:

  1. M-component (IgG or IgA) with persistent measurable paraprotein, or >=2 g monoclonal protein in 24 hr urine specimen or patients with an abnormal serum kappa/lambda ratio and a level of kappa or lambda light chain > 10 mg/dl.
  2. >=90 days and <= 120 days post transplant
  3. Laboratory values less than or equal to 2 weeks prior to initiation of treatment:

     * Absolute neutrophil count (ANC) greater than or equal 1.5 x 10^9/L
     * Platelets (PLT) greater than or equal to 100 x 10^9/L
     * Hemoglobin (Hgb) greater than or equal to 9 g/dL
     * Serum creatinine less than or equal to 1.5 upper limit of normal (ULN)
     * Serum bilirubin less than or equal to 1.5 ULN
     * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) less than or equal to 3.0 x ULN
     * Negative for proteinuria based on dip stick reading OR, if documentation of +1 result for protein on dip stick reading, then total urinary albumin ≤ 500 mg and measured creatinine clearance (CrCl) greater than or equal to 50 mL/min from a 24-hour urine collection
  4. A negative pregnancy test 48 hours prior to study treatment and must not be lactating if they are females of childbearing age.
  5. Ability to understand and the willingness to sign a written informed consent document in accordance with the guidelines of the Washington University Human Studies Committee.
  6. Age greater than or equal to 18 years old.
  7. ECOG performance status less than or equal to 2.

Exclusion Criteria:

1. Receiving any other investigational agents.
2. Receiving concurrent steroids with a dose equivalent of prednisone of >= 150 mg/month.
3. Female patients who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control. Barrier contraceptives must be used throughout the trial in both sexes. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study.
4. Biopsy proven amyloidosis.
5. Patients with a history of another primary malignancy within less than or equal to 5 years, with the exception of inactive basal or squamous cell carcinoma of the skin.
6. Prior chemotherapy less than or equal to 3 weeks prior to registration and/or randomization. Patients must have recovered from all therapy-related toxicities.
7. Prior biologic or immunotherapy less than or equal to 2 weeks prior to registration and/or randomization. Patients must have recovered from all therapy-related toxicities.
8. Prior full field radiotherapy less than or equal to 4 weeks or limited field radiotherapy less than or equal to 2 weeks prior to randomization. Patients must have recovered from all therapy-related toxicities.
9. Pleural effusion or ascites that cause respiratory compromise (greater than or equal to CTC grade 2 dyspnea).
10. Major surgery (i.e. laparotomy) less than or equal to 4 weeks prior to randomization. Minor surgery less than or equal to 2 weeks prior to randomization. Insertion of a vascular access device is not considered major or minor surgery in this regard. Patients must have recovered from all surgery-related toxicities.
11. Patients who have received investigational drugs less than or equal to 4 weeks prior to registration and/or randomization.
12. Prior therapy with anti-vascular endothelial growth factor (VEGF) agents.
13. Any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study:

    * Uncontrolled high blood pressure, history of labile hypertension, or history of poor compliance with an antihypertensive regimen
    * Unstable angina pectoris
    * Symptomatic congestive heart failure
    * Myocardial infarction less than or equal to 6 months prior to registration and/or randomization
    * Serious uncontrolled cardiac arrhythmia
    * QTc interval > 450 milliseconds in males or > 470 milliseconds in females Uncontrolled diabetes
    * Active or uncontrolled infection
    * Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
14. Acute or chronic liver disease (e.g. hepatitis, cirrhosis).
15. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PTK787/ZK 222584 (i.e., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, bowel obstruction, or inability to swallow the tablets).
16. Patients with confirmed diagnosis of human immunodeficiency virus (HIV) infection are excluded at the investigator's discretion if he/she feels that: a potential drug interaction between PTK787/ZK 222584 and any of the patient's anti-HIV medications could influence the efficacy of the anti-HIV medication, or it may place the patient at risk due to the pharmacologic activity of PTK787/ZK 222584.
17. Patients who are taking therapeutic warfarin sodium (Coumadin) or similar oral anticoagulants that are metabolized by the cytochrome P450 system. Heparin is allowed.
18. Patients unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 09/21/2005 and closed to participant enrollment on 06/17/2008.
Period: Overall Study
Arm/Group | PTK787/ZK 222584
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PTK787/ZK 222584
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 57 [38 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 21
Durie-Salmon stage at study entry [Number; unit: participants] — * Stage I:Hemoglobin (hgb) level >10.5 g/dL & calcium level is normal or ≤12 mg/dL & Low M-protein levels (IgG level is <5 g/dL; IgA level <3 g/dL) & Urine light chains <4 g per 24 hours, & Bone X-ray normal bone structure or a solitary bone plasmacytoma
  * Stage IIA:Levels of hgb, calcium, M-protein and Bence Jones protein fall somewhere between stages I and III & No kidney failure (creatinine ≤2 mg/dL)
  * Stage III: High M protein (IgG is>7 g/dL; IgA is >5g/dL) & Urine light chains >12 g per 24 hours & hgb <8.5 g/dL & calcium >2 m/dL) & X-ray studies of bone >3 lytic bone lesions
  participants
    Stage IA | 7
    Stage IIA | 7
    Stage IIIA | 7
International Staging System (ISS) at study entry [Number; unit: participants] — * Stage I:Beta 2-microglobulin level <3.5 mg/L & Albumin level ≥3.5 g/dL
  * Stage II Beta 2-microglobulin level <3.5 g/L & Albumin level <3.5 g/dL OR Beta 2-microglobulin level is 3.5 to 5.5 mg/L
  * Stage III Beta 2-microglobulin level is ≥5.5 mg/L
  participants
    Stage I | 17
    Stage II | 3
    Stage III | 1
Beta-2 Microglobulin at study entry [Median (Full Range); unit: mg/L] | 2.3 [1.2 to 5.65]
Paraprotein at study entry [Number; unit: participants]
  IgG | 18
  IgA | 3
Serum M-spike at study entry [Median (Full Range); unit: g/dL] | 0.5 [0 to 2.4]
Bone marrow aspirate plasma [Median (Full Range); unit: percentage of cells at study entry] | 5 [0 to 15]
Conventional cytogenetics [Number; unit: participants]
  Normal karyotype | 8
  Monosomy 13 | 1
  Hypodiploid karyotype with t(11;14) | 1
  Monosomy 13 and t(4:14) | 2
  Others | 8
  No available cytogenetics | 1

OUTCOME MEASURES:

1. Primary Outcome: Detectable Paraprotein Level (IgG or IgA)at ≤5 g/dL Who Show a 50% Reduction (Complete Response + Partial Response) in Their Paraprotein After Starting Treatment With the Study Drug
Time Frame: Day 90
Population: Participants were evaluable for response if they completed 3 cycles of treatment. 10 out of 21 participants completed 3 cycles of treatment.
Measure: Number; unit: participants
Arm/Group | PTK787/ZK 222584
Number analyzed (Participants) | 10
participants
  Complete response | 0
  Partial response | 1
  No response | 9

2. Secondary Outcome: Time to Progression
Description: Time to progression is from the start of treatment until the first date that criteria for progressive disease (PD) are met.
  * 25% increase in the level of the serum monoclonal paraprotein, which must also be an absolute increase of at least 0.5 g/dL and confirmed by at lease 1 repeated investigation.
  * 25% increase in the 24 hr urinary light chain excretion, which must also be an absolute increase of at least 200 mg/ 24 hr and confirmed by at least 1 repeated investigation.
  * 35% increase in plasma cells in a bone marrow aspirate or on trephine biopsy, which must also be an absolute increase of at least 10%.
    * Increase in the size of existing bone lesions or soft tissue plasmacytomas
    * New lytic bone lesions or soft tissue plasmacytomas or definite increase in the size of residual bone lesions (development of a compression fracture does not exclude continued response and may not indicate progression).
    * Hypercalcemia - corrected serum calcium > 11.5 mg/dL
Time Frame: Until the patient progresses or expires (up to 457 days)
Population: Participants were evaluable for time to progression if they completed 3 cycles of treatment. 10 out of 21 participants completed 3 cycles of treatment.
Measure: Median (Full Range); unit: days
Arm/Group | PTK787/ZK 222584
Number analyzed (Participants) | 10
days | 149 [28 to 457]

3. Secondary Outcome: Safety and Tolerability of PTK787/ZK 222584
Description: Number of Grade 3/4 adverse events per the National Cancer Institute (NCI) Common Toxicity Criteria v 3.0.
Time Frame: 30 days after treatment ends [median of 15 cycles (11-32)]
Population: Only 13 out of the 21 participants experienced a grade 3 or 4 adverse event.
Measure: Number; unit: adverse events
Arm/Group | PTK787/ZK 222584
Number analyzed (Participants) | 21
adverse events
  Gastrointestinal toxicity | 8
  Neurologic toxicity | 5
  Cardiac toxicity | 4
  Hematological toxicity | 3

4. Secondary Outcome: Disease Free Survival
Time Frame: Until the patient expires
Population: This secondary outcome was not analyzed.
Arm/Group | PTK787/ZK 222584
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of treatment up through 30 days following the end of treatment.
Arm/Group | PTK787/ZK 222584
Serious Adverse Events (participants affected / at risk) | 3/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PTK787/ZK 222584 (N=21)
Hypertension (Cardiac disorders) | 1
Infection without neutropenia (pneumonia) (Infections and infestations) | 1
Hypotension (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PTK787/ZK 222584 (N=21)
Abdominal pain (Gastrointestinal disorders) | 2
Alkaline phosphatase (Investigations) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Belching (Gastrointestinal disorders) | 1
Bilateral lower extremity edema (General disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 1
Cardiac troponin (Cardiac disorders) | 1
Chest pain (Musculoskeletal and connective tissue disorders) | 1
Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Diaphoresis (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Distension (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 4
Dog bite (Injury, poisoning and procedural complications) | 1
Dysgeusia (Gastrointestinal disorders) | 1
Dyspepsia/heartburn (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Early satiety (Gastrointestinal disorders) | 1
Elevated creatinine (Investigations) | 4
Erythema (Skin and subcutaneous tissue disorders) | 1
Facial flushing (Vascular disorders) | 1
Fatigue (General disorders) | 12
Fever - no infection (General disorders) | 3
Flatulence (Gastrointestinal disorders) | 1
GERD (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Generalized pain (General disorders) | 1
Headache (Nervous system disorders) | 7
Hemoglobin (Blood and lymphatic system disorders) | 6
Hiatal hernia (Musculoskeletal and connective tissue disorders) | 1
Hip pain (Musculoskeletal and connective tissue disorders) | 1
Hypercalcemia (Investigations) | 4
Hypercholesterolemia (Investigations) | 1
Hyperkalemia (Investigations) | 1
Hypermagnesemia (Investigations) | 1
Hypernatremia (Investigations) | 1
Hypertension (Cardiac disorders) | 7
Hypertriglyceridemia (Investigations) | 1
Hypoalbuminemia (Investigations) | 2
Hypocalcemia (Investigations) | 2
Hyponatremia (Investigations) | 1
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Infection with unknown ANC (Infections and infestations) | 1
Infection without neutropenia (Infections and infestations) | 6
Insomnia (Psychiatric disorders) | 2
Left ventricular dysfunction (Cardiac disorders) | 1
Leukocytes (WBC) (Investigations) | 5
Lower extremity pain (Musculoskeletal and connective tissue disorders) | 2
Lymphopenia (Investigations) | 6
Mental haziness (Nervous system disorders) | 1
Mood alteration - anxiety (Psychiatric disorders) | 2
Mood alteration - depression (Psychiatric disorders) | 1
Motor neuropathy (Nervous system disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Nausea (Gastrointestinal disorders) | 14
Neutrophils (ANC) (Investigations) | 5
Oral thrush (Gastrointestinal disorders) | 1
Platelets (Investigations) | 6
Post-herpetic neuralgia (Nervous system disorders) | 1
Prolonged QTC (Cardiac disorders) | 2
Proteinuria (Renal and urinary disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Rigors (General disorders) | 2
SGOT (AST) (Investigations) | 5
SGPT (ALT) (Investigations) | 7
Sensory neuropathy (Nervous system disorders) | 4
Sinus tachycardia (Cardiac disorders) | 1
Substernal (xiphoid) pain (Musculoskeletal and connective tissue disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 9
Weakness (Musculoskeletal and connective tissue disorders) | 1
Weight loss (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
In November 2008, it was reported that the drug might have carcinogenic potential in animal models. At that time, the remaining three patients were taken off study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes